CLINICAL TRIAL: NCT04538807
Title: A Study for Electrodiagnostic Finding According to the Type of Lumbar Disc Herniation on MRI
Brief Title: EMG Finding According to the Type of Lumbar Disc Herniation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yeungnam University Hospital (Other)
Responsible Party: Principal Investigator, Dong Gyu Lee, Assistant professor, Yeungnam University Hospital
Other Study IDs: 2020-07-005-001
Record Dates: First submitted 2020-08-21; First posted 2020-09-04 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Intervertebral Disc Displacement; Electromyography
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Electromyography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lumbar disc herniation: Patients are complaining of lower extremity radiating pain due to lumbar disc herniation.
  Interventions: Diagnostic Test: electromyography

INTERVENTIONS:
Diagnostic Test: electromyography — Electromyography (EMG) is an electrodiagnostic medicine technique for evaluating and recording the electrical activity produced by skeletal muscles.

SUMMARY:
Disc herniation is a common cause of low back pain and leg pain. Electromyography is the only test that can objectively examine nerve damage caused by a lumbar disc herniation. This study aimed to compare the MRI findings of disc herniation and the aspects of electromyography.

ELIGIBILITY:
Inclusion Criteria:

* Radicular pain within 6 months
* Disc herniation confirmed by lumbar MRI
* undergoing electromyography

Exclusion Criteria:

* Patients who refused electromyography
* Patients taking warfarin
* Lower limb amputation patient
* Pregnant women
* Patients who have undergone surgical treatment for disc herniation
* Patients with peripheral neuropathy ( AIDP, CIDP, diabetic amyotrophy, peroneal pals et al.)

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary referral hospital
Sampling Method: Non-Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Denervation pattern of muscles in lower extremity | 1 day During the examination of Electromyogram
  The location of the lower limb muscles where spontaneous activity occurs

SECONDARY OUTCOMES:
Disc herniation findings of lumbar MRI | 1 day During the examination of lumbar MRI
  Anatomical location of disc herniation

CONTACTS AND LOCATIONS:
Locations (1):
- Yeungnam University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No